CLINICAL TRIAL: NCT05480124
Title: Enhancing Neural Synchrony and Affective Cognitive Control in Bipolar Disorder Using Personalized Transcranial Alternating Current Stimulation (tACS)
Brief Title: Bipolar Transcranial Alternating Current Stimulation (tACS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Milken Institute (Other); Baszucki Brain Research Fund (Other)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00208557
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder
Keywords: transcranial alternating current stimulation (tACS); electroencephalogram (EEG)
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants, study coordinator, and clinical assessor will be blind as to which session the participants receive active or sham treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham stimulation treatment (Sham Comparator): Sham stimulation during a computerized task and electroencephalogram (EEG) recording.
  Interventions: Device: Sham stimulation treatment
- tACS brain stimulation treatment (Experimental): tACS brain stimulation during a computerized task and EEG recording. Participants will receive tACS using individualized peak Phase-amplitude coupling (PAC) frequency pairs determined in Session 1.
  Interventions: Device: tACS brain stimulation treatment

INTERVENTIONS:
Device: tACS brain stimulation treatment — Participants will wear an EEG cap on the head attached with EEG-recording and tACS electrodes. tACS will be delivered by passing a small electrical current via the tACS electrodes to the scalp to stimulate brain activity during a computerized behavioral task. The effect of active stimulation on EEG will be measured via EEG-recording electrodes during short rests (between stimulation blocks). The stimulation session will last for approximately 60 minutes. After treatment, participants will be asked about the experience and if there are any side effects.
  Arms: tACS brain stimulation treatment
Device: Sham stimulation treatment — Participants will wear an EEG cap on the head attached with EEG-recording and tACS electrodes. Sham tACS will be delivered by passing a transient (approximately 12 seconds ) small electrical current via the tACS electrodes during a computerized behavioral task. The effect of sham stimulation on EEG will be measured via EEG-recording electrodes during short rests (between stimulation blocks). The sham stimulation session will last for approximately 60 minutes. After treatment, participants will be asked about the experience and if there are any side effects.
  Arms: Sham stimulation treatment

SUMMARY:
The purpose of this clinical trial is to measure the safety and effectiveness of a non-invasive brain stimulation device called Transcranial Alternating Current Stimulation (tACS) in participants with bipolar disorder (BD).

Participants will be asked to come in for 3 sessions. If participants qualify at the screening visit (session 1) then enrolled participants will complete sessions 2 and 3 as well as have a 30-day follow-up phone call.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of BD based on Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria being met from previous enrollment in the Prechter Bipolar Longitudinal Study
* This study will select BD patients that scored above published norms (upper 50th percentile) on the NEO-PI impulsivity facet to ensure that the recruited patients exhibit the network dysfunction targeted by the tACS paradigm and therefore have the potential to benefit from this neuromodulation technique.
* Patients must be on a stable dose of medication for two weeks prior to Sessions 2 and 3.

Exclusion Criteria:

* Significant neurological abnormalities, such as seizure disorder, mass lesions, etc.
* Known Mendelian disorder
* Active problematic substance use in the past 30 days (as determined by the Substance Use Disorder module of SCID)
* Evidence of suicidal intentions or behaviors in the past month, as judged by affirmative responses to question number 4 or number 5 on the Columbia Suicide Severity Rating Scale (CSSRS) or report of suicidal behaviors in the last 6 months
* Pregnant or trying to become pregnant, or currently lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan F Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham First, Then tACS: Participants in this arm received the sham stimulation treatment during session 2 and then received the tACS brain stimulation treatment in session 3.
- tACS, Then Sham: Participants in this arm received the tACS brain stimulation treatment in session 2 and then received the sham stimulation treatment during session 3.
Period: Session 1 (Baseline)
Arm/Group | Sham First, Then tACS | tACS, Then Sham
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Session 2
Arm/Group | Sham First, Then tACS | tACS, Then Sham
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Washout
Arm/Group | Sham First, Then tACS | tACS, Then Sham
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0
Period: Session 3
Arm/Group | Sham First, Then tACS | tACS, Then Sham
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham First, Then tACS | tACS, Then Sham | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (10.03) | 42.75 (12.44) | 42.0 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 7 | 14
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Severity of Side Effects Reported at End of Stimulation Session as Reported by the Participant on the Stimulation Side Effects Questionnaire.
Description: The score was calculated by summing the severity score of items that were rated by the participant as related to stimulation on the Stimulation Side Effects Questionnaire. There was a total of 14 symptoms listed on the questionnaire. Participants rated each item rated on a scale of 0-4, with 0 meaning no relation and 4 meaning definitely related. The total possible range of the questionnaire was 0-56.
Time Frame: Up to 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
Number analyzed (Participants) | 18 | 18
score on a scale | 5.66 (4.47) | 5.00 (0.90)
Statistical Analysis 1: Comparison: Sham Stimulation Treatment vs tACS Brain Stimulation Treatment; Test type: Superiority; p = 0.609, t-test, 2 sided

2. Primary Outcome: Participants Who Withdrew During or After the Stimulation Session
Description: Results reflect the number of participants who withdrew from the trial during or after a stimulation session with either the tACS or the sham stimulation treatment.
Time Frame: Up to 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

3. Primary Outcome: Accuracy Signal Detection Theory Metric Sensitivity (d') Derived From the Behavioral Responses to Go and NoGo Trials on the Cognitive Control Task.
Description: The Go/NoGo task was a cognitive task, where participants were shown "go" stimuli (i.e., go trials) and "no-go" stimuli and responded by pressing a button when seeing "go" stimuli and not responding when seeing the "no-go" stimuli. Accuracy was measured by calculating D' (D prime), which provided a measure of perceptual sensitivity to the differing stimuli. Larger values of D' indicated greater discernability (i.e., accuracy) between the Go and NoGo trials. D-prime, also called the sensitivity index represents how well someone can detect a signal amidst background noise. At its core, D-prime is the standardized difference between the means of the Signal Present and Signal Absent distributions, which can be calculated by taking the difference between the Z-score of the False Alarm Rate and the Z-scores of the Hit Rate. A D-prime of 0 means no sensitivity. Negative D-prime values are rare and may indicate errors or reversed interpretations of hits and false alarms.
Time Frame: Up to 3 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
Number analyzed (Participants) | 18 | 18
z-score | 2.08 (0.51) | 2.20 (0.56)
Statistical Analysis 1: Comparison: Sham Stimulation Treatment vs tACS Brain Stimulation Treatment; Test type: Superiority; p = 0.098, t-test, 2 sided

4. Primary Outcome: Accuracy Signal Detection Theory Metric Response Bias Derived From the Behavioral Responses to Go and NoGo Trials on the Cognitive Control Task.
Description: The Go/NoGo task was a cognitive task, where participants were shown "go" stimuli (i.e., go trials) and "no-go" stimuli and responded by pressing a button when seeing "go" stimuli and not responding when seeing the "no-go" stimuli. Response bias was measured using beta, such that more negative beta values indicated a stronger tendency to respond to all stimuli, regardless of "go" or "no-go" status. Response bias is indexed by taking the average between the Z-score of the False Alarm Rate and the Z-scores of the Hit Rate. A higher response bias indicates that the participant is more likely to respond "signal absent" (favors avoiding false alarms but increases misses). A response bias of 0 means the individual equally weighs the costs of misses and false alarms. A more negative response bias indicated that the participant is more likely to respond "signal present" (favors hits but increases false alarms).
Time Frame: Up to 3 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
Number analyzed (Participants) | 18 | 18
z-score | -0.03 (0.28) | -0.05 (0.22)
Statistical Analysis 1: Comparison: Sham Stimulation Treatment vs tACS Brain Stimulation Treatment; Test type: Superiority; p = 0.204, t-test, 2 sided

5. Primary Outcome: Reaction Time (in Milliseconds) of Go Trials on the Cognitive Control Task
Description: Participants' reaction time to responding to the "Go" signal during the Go/NoGo task was measured.
Time Frame: Up to 3 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
Number analyzed (Participants) | 18 | 18
milliseconds | 584.88 (97.55) | 582.01 (88.98)
Statistical Analysis 1: Comparison: Sham Stimulation Treatment vs tACS Brain Stimulation Treatment; Test type: Superiority; p = 0.383, t-test, 2 sided

6. Primary Outcome: Theta-gamma Phase Amplitude Coupling (PAC) (Kullback-Leibler Modulation Index) During the Rest EEG Blocks Interleaved Between Stimulation Blocks.
Description: Theta-gamma phase-amplitude coupling (PAC) is a neural phenomenon observed in the brain, where the phase of slower theta oscillations modulates the amplitude of faster gamma oscillations. This type of coupling is thought to play a critical role in various cognitive control. For the trial, higher PAC values indicated higher levels of coupling or connection between the two frequencies (i.e., increased cognitive control).
Time Frame: Up to 3 weeks
Population: Data was not collected from 1 participant in the sham arm, as their EEG data was unreadable following administration of the sham.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
Number analyzed (Participants) | 17 | 18
arbitrary units | 0.14 (0.12) | 0.20 (0.32)
Statistical Analysis 1: Comparison: Sham Stimulation Treatment vs tACS Brain Stimulation Treatment; Test type: Superiority; p = 0.201, t-test, 2 sided

7. Other Pre Specified Outcome: Emotional Flanker Task - Accuracy
Description: After completing the Emotion Go-NoGo task, participants will complete another cognitive control task (i.e., Emotional Flanker Task) with gray-scaled unpleasant, pleasant, and neural images from the International Affective Picture System. Participants are tasked with indicating which valance is presented in certain images while ignoring other images. Accuracy is defined as the percentage of trials that the participant correctly reports the valance of the target image. The total number of correct trials will be divided by the total number of trials to obtain an accuracy score. Average accuracy scores per condition and total will be calculated.
Time Frame: Approximately 30-60 minutes after the Go-NoGo task at all three time points (baseline, session 1, session 2)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Emotional Flanker Task - Reaction Time
Description: Reaction time will also be collected during the Emotional Flanker Task. Reaction time is defined as the length of time it takes the participant to respond after the onset of the stimuli. Average reaction times per condition and total will be calculated.
Time Frame: Approximately 30-60 minutes after the Go-NoGo task at all three time points (baseline, session 1, session 2).
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Emotional Flanker Task - EEG
Description: EEG will also be collected during the Emotional Flanker Task. Phase-amplitude coupling will be calculated and defined as the coupling between the amplitude of high frequency oscillations (e.g., gamma) and low frequency phase (e.g., theta). Average coupling scores per condition and total will be calculated.
Time Frame: Approximately 30-60 minutes after the Go-NoGo task at all three time points (baseline, session 1, session 2).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 7 weeks
Description: Participants were called 30 days after the final visit and asked if they had any side effects from the tACS.
Arm/Group | Sham Stimulation Treatment | tACS Brain Stimulation Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT05480124/Prot_SAP_000.pdf